CLINICAL TRIAL: NCT02576249
Title: Does Anesthetic Contribute to Symptomatic Relief in Corticosteroid Injections for Knee Osteoarthritis? A Double-Blind Randomized Trial Comparing Corticosteroid/Ropivacaine Versus Corticosteroid/Saline Injections
Brief Title: Corticosteroid/Ropivacaine Versus Corticosteroid/Saline Injections for Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jacob L. Sellon, M.D., Assistant Professor of Physical Medicine and Rehabilitation, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-003120
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; injection; steroid; anesthetic
MeSH Terms: conditions — Osteoarthritis | interventions — Ropivacaine; Saline Solution; Sodium Chloride; Methylprednisolone; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ropivacaine and Methylprednisolone (Active Comparator): 0.2% ropivacaine and methylprednisolone knee joint injection
  Interventions: Drug: Ropivacaine; Drug: Methylprednisolone
- Saline and Methylprednisolone (Experimental): 0.9% normal saline and methylprednisolone knee joint injection
  Interventions: Drug: Normal saline; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Ropivacaine — 4cc 0.5% ropivacaine
  Other Names: Naropin
  Arms: Ropivacaine and Methylprednisolone
Drug: Normal saline — 4cc of sterile normal saline (0.9%)
  Other Names: Sodium Chloride
  Arms: Saline and Methylprednisolone
Drug: Methylprednisolone — 1cc 40mg methylprednisolone
  Other Names: Depo-Medrol

SUMMARY:
Corticosteroid injections are commonly used for the symptomatic treatment of knee osteoarthritis. Common practice is to inject the joint with a combination of corticosteroid and local anesthetic, with the rationale of providing longer duration pain relief with the corticosteroid and immediate, though short duration relief with the anesthetic. However, multiple in vitro and animal studies have shown that local anesthetic may be harmful to chondrocytes. Despite this data, use of intra-articular anesthetic remains widespread. Many clinicians believe incorporating the anesthetic is important because it can provide immediate pain relief and facilitate patient confidence in the treatment program. However, there is no published data to validate this reasoning. Therefore, the anesthetic has unknown clinical benefit and may have adverse effects on articular cartilage. In light of this, the investigators question the routine use of anesthetics in joint injections. The purpose of this study is to compare the effects of knee joint injections using: 1) corticosteroid with local anesthetic versus 2) corticosteroid with normal saline.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 or older
2. Knee osteoarthritis (uni- or bilateral) as defined by the American College of Rheumatology (staged by Kellgren-Lawrence radiographic grading scale)

Exclusion criteria:

1. Rheumatologic/inflammatory disease
2. Metabolic bone disease
3. Crystalline arthropathy
4. Current smoking
5. BMI > 40
6. Knee injection with corticosteroid or viscosupplementation within previous 6 months
7. History of knee prolotherapy, platelet rich plasma or cellular (stem cell) injection
8. Knee surgery within the last year
9. Chronic opioid use
10. Chronic pain syndrome/fibromyalgia
11. Pain behavior during the clinical encounter as judged by the injecting physician
12. Physician specifically ordered injection of corticosteroid/anesthetic or other specific combined corticosteroid injection
13. Diagnostic uncertainty by referring provider
14. Referral for bilateral knee or multiple joint injections (*note that arthritis involving multiple joints alone is not an exclusion criteria, only the patient receiving more than 1 injection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob L Sellon, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine and Methylprednisolone | Saline and Methylprednisolone
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine and Methylprednisolone | Saline and Methylprednisolone | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (7.43) | 57 (11.8) | 57 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 7 | 6 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 29
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (7.68) | 30.9 (6.46) | 30.4 (7.01)
Knee Effusion [Count of Participants; unit: Participants] — Knee effusion, colloquially known as water on the knee, occurs when excess fluid accumulates in or around the knee joint.
  Participants
    Yes | 5 | 4 | 9
    No | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Knee Osteoarthritis Outcome Score (KOOS) Pain Subscale
Description: The KOOS holds 42 items in five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Time Frame: 3 months after the injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropivacaine and Methylprednisolone | Saline and Methylprednisolone
Number analyzed (Participants) | 15 | 14
units on a scale | 63.1 (16.1) | 67.2 (14.4)

2. Secondary Outcome: Pain Scale Score
Description: Pain was measured by a Visual Analog Scale (VAS) marked from 0 (no pain) to 10 (unbearable pain) at rest and with activity. It was collected at baseline (pre-injection), immediately post-injection on the day of surgery, and at 2 weeks and 3 months.
Time Frame: Pre-injection, immediately post-injection, 2 weeks, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropivacaine and Methylprednisolone | Saline and Methylprednisolone
Number analyzed (Participants) | 15 | 14
units on a scale
  Pre-injection Activity | 6.4 (2) | 5.8 (2.5)
  Pre-injection Rest | 2.4 (2) | 4 (2)
  Immediately Post-injection Activity | 1.9 (2.3) | 2.4 (2.2)
  Immediately Post-injection Rest | 1.2 (1.5) | 1.4 (1.7)
  2 Weeks Activity | 3.6 (2.5) | 3.6 (2)
  2 Weeks Rest | 1.7 (2) | 2.7 (2.2)
  3 Months Activity | 3.9 (2.7) | 4.6 (2.4)
  3 Months Rest | 2.6 (2.2) | 2.8 (2.4)

3. Secondary Outcome: Tegner Activity Level Scale
Description: The Tegner activity level scale is a scale that aims to provide a standardized method of grading work and sporting activities. The Tegner activity level scale is a graduated list of activities of daily living, recreation, and competitive sports. The patient is asked to select the level of participation that best describes their current level of activity and that before injury.
  A score of 0 represents sick leave or disability pension because of knee problems, whereas a score of 10 corresponds to participation in national and international elite competitive sports. A score >6 can only be achieved if the person participates in recreational or competitive sport.
Time Frame: baseline (pre-injection), 2 weeks, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropivacaine and Methylprednisolone | Saline and Methylprednisolone
Number analyzed (Participants) | 15 | 14
units on a scale
  baseline (pre-injection) | 3.5 (2.2) | 3.0 (1.6)
  2 weeks | 4.3 (1.7) | 3.2 (1.3)
  3 months | 3.5 (2.1) | 3 (1.7)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Ropivacaine and Methylprednisolone | Saline and Methylprednisolone
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

LIMITATIONS AND CAVEATS:
Lack of power due to lower than expected enrollment; follow-up was limited to 3 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes